CLINICAL TRIAL: NCT03999294
Title: The Influence of the Bmgim Music Therapy Method in the Reduction of Stress in Patients With Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis): Quantitative and Qualitative Study
Brief Title: Bmgim Music Therapy Method in Reducing Stress in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universidad Católica de Valencia San Vicente Mártir (Unknown); Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Vicente J Prado Gascó, Profesor Ayudante Doctor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: musicoterapia25f2015
Record Dates: First submitted 2019-06-05; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Bowel Diseases, Inflammatory; Crohn Disease; Colitis, Ulcerative
Keywords: Music Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Experimental Group (Experimental)
  Interventions: Other: BMGIM Music Therapy Method

INTERVENTIONS:
Other: BMGIM Music Therapy Method — The BMGIM method is today one of the models recognized by the international music therapy community, deserving this distinction those approaches that develop a solid theoretical and practical body, with specific training programs as training for new therapists, and that also promote the scientific research as a way to develop the method and Music Therapy.
  Arms: Experimental Group

SUMMARY:
Inflammatory bowel disease (IBD) is a term that defines a chronic disease characterized by inflammation of the intestine. It includes ulcerative colitis (UC) and Crohn's disease (CD). The objective of the study was to administer a treatment based on a group adaptation of the BMGIM in patients with inflammatory bowel disease (IBD) and assess its impact on state of mind, quality of life, anxiety, depression, immunocompetence as a marker of well-being, and levels of acute and chronic stress.

To achieve the objectives a quasi-experimental, quantitative, qualitative, analytical, and prospective study was performed. 41 patients with IBD divided into a test group (24 patients), who received 8 sessions over 8 weeks, and a control group (17 patients). A saliva sample was taken from each patient before and after each session to determine cortisol levels (acute stress) and IgA (immunocompetence) using ELISA. A series of questionnaires were completed as follows: HADS (perceived anxiety), MOOD (state of mind), and CCVEII (quality of life). Similarly, a hair sample was taken before the first and after the last session to determine the cumulative cortisol level (chronic stress) using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Diagnosed IBD (EC or UC) in the remission phase,
* They did not receive treatment with corticosteroids at least in the two months prior to the start of the study,
* They did not receive any extra pharmacological treatment,
* Attend the collaborating hospital center with the study, in this case, the University General Hospital of Valencia,
* Attend the schedule and schedule established for the study,
* Accept the conditions of participation in the study indicated in the signed informed consent prior to the start of the study
* * Do not take corticosteroids during the 8 weeks between the pre-test and the post-test,
* * Perform the pre-test before starting session 1 (in case of experimental group) or appointment 1 (in case of control group); and then the retest at the end of session 8 (in the case of an experimental group) or appointment with nursing after 8 weeks (in the case of a control group).
* * In the case of the patients belonging to the experimental group, who at the end of the 8 weeks of treatment would have attended at least 6 of the 8 sessions established (and that, obligatorily, 2 of them were 1 and 8, where the shots were taken) sample and completed the questionnaires).

Exclusion Criteria:

The patients who were excluded from this study were those who did not meet the requirements indicated in the inclusion criteria, or who showed aversion or rejection to this type of therapy.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Change in biological markers in saliva samples using enzyme-linked immunosorbent biological markers assay (ELISA) (PRE and POST Measures). | Baseline up to 8 weeks of treatment
  Quantifying change in biological markers in saliva samples using enzyme-linked immunosorbent assay (ELISA). (IgA level & Salivary Cortisol) comparing pre and post intervention
Change in biological markers in hair using enzyme-linked immunosorbent assay (ELISA).(PRE and POST Measures). | Baseline up to 8 weeks of treatment
  Quantifying change in biological markers in hair (Cortisol Hair) comparing pre and post intervention
Change in Hospital Anxiety and Depression Scale (HADS) (PRE and POST Measures) | Baseline up to 8 weeks of treatment
  14 items. 7 items for Anxiety and 7 for Depression. The score for the items is evaluated on a Likert scale ranging from 0 to 3 points, where 0 represents never or almost never, 1 a little or from time to time, 2 somewhat less than before or not as intense, and 3 maximum or almost always. Lastly, it is worth mentioning that these scales are interpreted based on the sum of each dimension, with 21 as the maximum, both for depression and for anxiety. Higher values represent a worse outcome. Observing change comparing pre and post intervention
Change in Short-form Questionnaire on Quality of Life in IBD (CCVEII-9) (PRE and POST Measures) | Baseline up to 8 weeks of treatment
  9 items grouped in a single dimension The final score is expressed on a scale of 0 to 100 points, such that a lower score corresponds to a lower quality of life and vice versa. Observing change comparing pre and post intervention
Change in the MOOD questionnaire (PRE and POST Measures). | Baseline up to 8 weeks of treatment
  The scale evaluates the frequency of the different states of mind (happiness, anger, sadness, and fear) based on 20 items (4 dimensions of 5 items each). The responses for the items were measured using a 3-point Likert scale (1=never, 2=sometimes, 3=often). Each dimension range from 1 to 3. There is not a total of all dimensions together. a lower score corresponds to high level fo that mood (lower values= a betwer outcome on anger, sadness, and fear and worst outcome on hapiness). Observing change comparing pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Javier Prado Gascó, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03999294/Prot_SAP_000.pdf